CLINICAL TRIAL: NCT04033809
Title: Effectiveness of High Fiber Multigrain Supplementation Among the Rheumatoid Arthritis Patients: A Randomized, Open Label Trial
Brief Title: Effectiveness of Multigrain Supplementation Among the Rheumatoid Arthritis Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universiti Sains Malaysia (Other)
Responsible Party: Principal Investigator, Dr. Lee Lai Kuan, Principal Investigator, Universiti Sains Malaysia
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: USM/JEPeM/19010081
Record Dates: First submitted 2019-07-16; First posted 2019-07-26 (Actual); Last update posted 2023-05-10 (Actual); Status verified 2023-05

CONDITIONS: Rheumatoid Arthritis
Keywords: Rheumatoid Arthritis; Fiber; Multigrain
MeSH Terms: conditions — Arthritis, Rheumatoid

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Multigrain powder (S) (Active Comparator): Oral high fiber multigrain supplements
  Interventions: Dietary Supplement: Multigrain powder (S)
- Standard care (C) (No Intervention): Standard care without oral high fiber multigrain supplements

INTERVENTIONS:
Dietary Supplement: Multigrain powder (S) — A twice daily high fiber multigrain powder supplementation for 12 weeks
  Arms: Multigrain powder (S)

SUMMARY:
The objective of this study is to evaluate the effect of high fiber multigrain supplementation on the level of clinical disease severity measures, blood inflammatory molecules, and nutritional status changes in RA patients.

DETAILED DESCRIPTION:
Rheumatoid Arthritis (RA) is a chronic inflammatory, autoimmune rheumatic disease, resulting in progressive joint inflammation and destruction. At present, there is no known cure for this disease. As a consequence of the potential side effects, many RA patients turn to other alternative remedies such as specialised diets and/or dietary supplements in a bid to relieve their symptoms. Therefore, the current study aims to examine the effectiveness of high fiber multigrain supplementation on the level of clinical disease severity measures, blood inflammatory molecules, together with the nutritional status changes in RA patients, as compare with conventional drug treatments.

ELIGIBILITY:
Inclusion Criteria:

* RA patients according to the American College of Rheumatology (ACR)
* Moderate (DAS 28 = 3.2 - 5.1) and severe (DAS 28 > 5.1) RA manifestation
* Chronological age: 21 years and above
* Stable RA patients who are receiving NSAIDs, glucocorticoids/DMARDs (for example leflunomide, methotrexate, sulfasalazine and hydroxychloroquine) for at least 3 months prior to entering the study
* Not taking antioxidant/antiinflammatory supplements (Example of antioxidant: vitamin C, vitamin E, grape seed extract, garlic capsule, ginkgo biloba) (Example of anti-inflammatory supplement: fish oil, curcumin extract, ginger extract, spirulina)

Exclusion Criteria:

* Having liver (chronic liver failure, cirrhosis, all types of hepatitis), kidney (chronic kidney disease, haemodialysis) or haematological (anaemia, thalassemia, haemophilia) disorders
* Active gastric/duodenal ulcer
* Psychiatric disease/mental retardation (bipolar disorder, depression, schizophrenia)
* Cancer (all types), Diabetes Mellitus (Type I and II), uncontrolled hypertension (BP at 140/90 mmHg for the past 3 months), and endocrine disorders (Cushing's disease, gigantism and hyperthyroidism).
* Alcohol and drug abuse (self-mentioned or as recorded in the medical card)
* Other autoimmune/inflammatory diseases (systemic lupus erythematosus, multiple sclerosis, gout, psoriasis, chronic inflammatory demyelinating polyneuropathy)
* Pregnancy/lactation
* Hormone replacement therapy (for at least 3 months prior to entering the study)
* Herbal remedies (any parts from the plants such as flowers, rhizome, seeds, roots, leaves, fruits, stems)
* Vegetarian patient (pure vegan)
* Gluten intolerance
* Participations from another supplementary program

Ages: 21 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 54 (Actual)
Dates: Start 2019-05-30 (Actual); Primary Completion 2019-09-30 (Actual); Study Completion 2019-12-31 (Actual)

PRIMARY OUTCOMES:
Disease Activity Score-28 (DAS-28) | Baseline and 12 weeks
  The DAS-28 is a system developed and validated by the EULAR (European League Against Rheumatism) to measure the progress and improvement of Rheumatoid Arthritis. DAS-28 values range from 2.0 to 10.0, while higher values mean a higher disease activity. The complex mathematical calculation is calculated by incorporating the value of erythrocyte sedimentation rate (ESR) and Visual Analog Scale (VAS). ESR (mm/hr) determines the severity of inflammatory response and monitor the effect of treatment. VAS is an indicator for pain intensity and patient global health, and the following cut points have been recommended: no pain (0-4 mm), mild pain (5-44 mm), moderate pain (45-74 mm), and severe pain (75- 100 mm).
  DAS-28 = 0.56 * sqrt(tender28) + 0.28 * sqrt(swollen28) + 0.70 * ln(ESR) + 0.014 * GH
  The scale categorises RA manifestations as mild (DAS-28: <3.2), moderate (DAS-28: 3.2-5.1) or severe (DAS-28: >5.1)
Health Assessment Questionnaire-Disability Index (HAQ-DI) | Baseline and 12 weeks
  The HAQ-DI is used to measure physical functionality. The HAQ-DI is usually analyzed by calculating scores. The single scales range from 0 (no difficulty) to 3 (unable to do). The total score ranges from 0-24, and higher score indicates severe disability.

SECONDARY OUTCOMES:
Blood glucose level | Baseline and 12 weeks
  Blood glucose is measured in mmol/L
Glycated hemoglobin (HbA1c) | Baseline and 12 weeks
  Glycated hemoglobin (HbA1c) is measured in %
White blood cell (WBC) count | Baseline and 12 weeks
  White blood cell (WBC) differential count is measured in x10^9/L
Red blood cell (RBC) count | Baseline and 12 weeks
  Red blood cell (RBC) count is measured in x10^12/L
Hemoglobin (Hb) | Baseline and 12 weeks
  Hemoglobin (Hb) is measured in g/dl
Hematocrit (Hct) | Baseline and 12 weeks
  Hematocrit (Hct) is measured in %
Mean corpuscular volume (MCV) | Baseline and 12 weeks
  Mean corpuscular volume (MCV) is measured in l/cell
Mean corpuscular hemoglobin (MCH) | Baseline and 12 weeks
  Mean corpuscular hemoglobin (MCH) is measured in g/cell
Platelet (PLT) count | Baseline and 12 weeks
  Platelet (PLT) count is measured in x10^9/L
Total cholesterol | Baseline and 12 weeks
  Total cholesterol is measured in mmol/L
Low density lipoprotein (LDL)-cholesterol | Baseline and 12 weeks
  Low density lipoprotein (LDL)-cholesterol is measured in mmol/L
High density lipoprotein (HDL)-cholesterol | Baseline and 12 weeks
  High density lipoprotein (HDL)-cholesterol is measured in mmol/L
Triglyceride (Tg) | Baseline and 12 weeks
  Triglyceride (Tg) is measured in mmol/L
Sodium level | Baseline and 12 weeks
  Sodium level is measured in mmol/L
Potassium level | Baseline and 12 weeks
  Potassium level is measured in mmol/L
Chloride level | Baseline and 12 weeks
  Chloride level is measured in mmol/L
Blood urea nitrogen (BUN) level | Baseline and 12 weeks
  Blood urea nitrogen (BUN) level is measured in mmol/L
Serum creatinine level | Baseline and 12 weeks
  Serum creatinine level is measured in umol/L
Calcium level | Baseline and 12 weeks
  Calcium level is measured in mmol/L
Uric acid level | Baseline and 12 weeks
  Uric acid level is measured in umol/L
Phosphorus level | Baseline and 12 weeks
  Phosphorus level is measured in mmol/L
Albumin | Baseline and 12 weeks
  Albumin is measured in g/L
Total protein | Baseline and 12 weeks
  Total protein is measured in g/L
Total bilirubin | Baseline and 12 weeks
  Total bilirubin is measured in umol/L
Alkaline phosphatase (ALP) | Baseline and 12 weeks
  Alkaline phosphatase (ALP) is measured in U/L
Alanine transaminase (ALT) | Baseline and 12 weeks
  Alanine transaminase (ALT) is measured in U/L
Aspartate transaminase (AST) | Baseline and 12 weeks
  Aspartate transaminase (AST) is measured in U/L
Serum interleukin-6 (IL-6) | Baseline and 12 weeks
  Interleukin-6 (IL-6) is a pleiotropic cytokine with a pivotal role in the pathophysiology of rheumatoid arthritis. The level correlates with the disease activity and joint destruction. Serum IL-6 is measured in pg/ml
Serum interleukin 1β (IL-1β) | Baseline and 12 weeks
  Interleukin 1β is among the most important proinﬂammatory cytokines in rheumatoid arthritis. Serum IL-1β is measured in pg/ml
Tumor necrosis factor-alpha (TNF-α) | Baseline and 12 weeks
  Tumor necrosis factor-alpha (TNF-α) is a proinflammatory cytokine that plays a pivotal role in regulating the inflammatory response in rheumatoid arthritis. Serum IL-1β is measured in pg/ml
High sensitivity-C-Reactive Protein (hs-CRP) | Baseline and 12 weeks
  High sensitivity-C-Reactive Protein (hs-CRP) is a disease activity marker in rheumatoid arthritis. Serum hs-CRP is measured in pg/ml
Serum matrix metalloproteinase-3 (MMP-3) | Baseline and 12 weeks
  MMP-3 is increased in rheumatoid arthritis, and has been proposed as a marker of joint damage and systemic inflammation. Serum MMP-3 is measured in ng/ml
Body mass index (BMI) | 12 weeks
  Body weight (in kilograms) and standing height (in meters) will be measured to indicate nutritional status. The weight and height will be combined to report BMI in kg/m^2
Waist hip ratio | 12 weeks
  Waist (in cm) and hip (in cm) circumferences will be measured to indicate obesity. This is calculated as waist measurement divided by hip measurement.
Body fat | Baseline and 12 weeks
  Body fat is measured in %
Fat mass | Baseline and 12 weeks
  Fat mass is measured in %
Fat free mass | Baseline and 12 weeks
  Fat free mass is measured in %
Total body water | Baseline and 12 weeks
  Total body water is measured in L
Estimated average required energy | Baseline and 12 weeks
  Estimated average required energy is measured in kcal
Tolerability assessment | At 4 weeks, 8 weeks and 12 weeks
  The participant's complaints of gastrointestinal discomfort upon supplement consumption such as heart burn, diarrhea, nausea, vomiting and headache will be recorded, and it will be reported as the frequency (n) of discomfort episodes.
Compliance assessment | At 4 weeks, 8 weeks and 12 weeks
  Remaining sachet counting: The remaining sachet/unfinished sachet will be counted, and compliance will be reported as %.

CONTACTS AND LOCATIONS:
Overall Officials: Lai Kuan Lee, PhD, Principal Investigator — Universiti Sains Malaysia
Locations (1):
- Universiti Sains Malaysia, Kubang Kerian, Kelantan, Malaysia

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-05-30): https://cdn.clinicaltrials.gov/large-docs/09/NCT04033809/Prot_SAP_000.pdf